CLINICAL TRIAL: NCT01580332
Title: NON-INVASIVE BIOMARKERS FOR EARLY DETECTION OF LUNG CANCERS: ELEMENT 1: NON-RANDOMIZED PHASE II EVALUATION AND VALIDATION IN NEWLY DIAGNOSED LUNG CANCER PATIENTS
Brief Title: Non-Invasive Biomarkers For Early Detection Of Lung Cancers
Acronym: ISRUSAL01
Status: Completed | Type: Observational
Sponsor: Douglas W. Johnson MD, FACR (Other)
Responsible Party: Sponsor-Investigator, Douglas W. Johnson MD, FACR, Principal Investigator, Baptist Cancer Institute
Organization: Baptist Cancer Institute (Other)
Other Study IDs: ISRUSAL01
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2012-04

CONDITIONS: Lung Cancer
Keywords: biomarkers; lung cancer; solitary pulmonary nodules; SPN; breath analysis; VOC; volatile organic compounds; sputum; auto-antibodies
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum; sputum
Oversight: Data Monitoring Committee: No

SUMMARY:
Recent studies have shown that low-dose chest CT scans can detect lung cancers in high-risk populations (age >50yo, >30 pack-years of tobacco use), and can lower cancer mortality. Unfortunately, the vast majority of "positive" findings on these CT scans are benign (>95%). Currently, an inordinate amount of expensive follow-up testing is required for these patients to try to prove who among them truly has a cancer.

Several new emerging non-invasive and potentially cheaper tests are now being investigated to help differentiate patients with cancers versus just benign lung nodules. These new tests include a new type of sputum analysis, a breath analysis, a blood test measuring certain tumor markers, a blood test looking for auto-antibodies, and a standard PET/CT scan. Each of these tests have different sensitivity and specificity rates when looking for lung cancer, and it is unclear which test is best.

This study will employ a panel of all 5 of these non-invasive tests on an initial cohort of 50 patients with recently diagnosed lung cancer to try to measure the sensitivity of the tests. A follow-on study will then perform the same panel of tests on 300 lung nodule patients to see which test, or combination of tests, gives the best overall accuracy in terms of predicting who really has lung cancer. It is hoped that the use of such a panel could lead to dramatically decreased need for expensive and morbid invasive testing for this population.

DETAILED DESCRIPTION:
The study revolves around specifying the exact signatures and accuracy associated with discriminating between benign and malignant SPNs for each of the biomarkers in the specific high risk cohort under the NLST screening protocol. To help identify and quantify these signatures, we will evaluate specifically the volatile signature in the exhaled breath, the accuracy of LuCED sputum detection, the profile of tumor markers and the specifications of auto-antibodies through immunoassays and Orbitrap technology, and the PET/CT in patients already diagnosed with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed cancer, prior to treatment

Exclusion Criteria:

* prior treatment for this cancer
* a history of any other cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient with newly diagnosed lung cancer (any histology, any stage) who has not yet begun definitive treatment, and who has no prior history of cancer of any type
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W Johnson, MD, Principal Investigator — Baptist Cancer Institute
Locations (1):
- Baptist Cancer Institute, Baptist Medical Center, Jacksonville, Florida, United States